CLINICAL TRIAL: NCT02712346
Title: The Role of Endothelin-1 in Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Gilead Sciences (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Abdullah Kutlar, Professor of Medicine, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Endothelin; 5U01HL117684 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2016-03-18 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle Cell Anemia; Sickle Cell Thalassemia; Sickle Beta Thalassemia; Proteinuria; Sickle nephropathy
MeSH Terms: conditions — Anemia, Sickle Cell; Proteinuria | interventions — ambrisentan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Ambrisentan 5 mg PO daily
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): One inactive pill PO daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan 5 milligrams a day or a placebo (sugar pill) for twelve weeks
  Other Names: Letairis
  Arms: Treatment
Drug: Placebo — One inactive pill daily for twelve weeks
  Other Names: "Sugar Pill"
  Arms: Placebo

SUMMARY:
The primary goal of the study is to determine the safety and tolerability of ambrisentan. It is also expected that ambrisentan will improve blood flow in the lungs, decrease inflammation, and reduce pain in sickle cell patients. An additional goal is to evaluate the use of select biomarkers in evaluating sickle nephropathy.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that endothelin antagonist (ETA) receptor blockade using ambrisentan is safe, tolerable, and improves kidney function/albuminuria in patients with sickle cell disease (SCD). The investigators anticipate a reduction in proteinuria, a decrease in tricuspid regurgitation jet (TRJ) velocity, reduction in inflammatory markers, improvement in forearm blood flow, and improvement in nociception/pain.

The primary efficacy endpoint was chosen as the effect of ETA receptor blockade on the reduction of microalbuminuria based upon findings in diabetic nephropathy, which has a similar pathogenesis to sickle nephropathy. A 30% reduction in proteinuria is rather conservative and realistic based upon the results of studies of ETA receptor blockade in diabetic nephropathy that consistently resulted in 40-45% reduction in proteinuria. Pre-clinical data has shown that changes can be detected in urinary nephrin excretion before overt proteinuria is observed in a model of chronic ET-1 elevation. Furthermore, tubular injury that can occur as a result of an intrarenal vaso-occlusive crisis (VOC) should be expected to increase the level of renal tubular injury markers, neutrophil gelantinase-associated lipocalin (NGAL), kidney injury molecule-1 (KIM-1), and netrin. Treatment with ambrisentan would be expected to attenuate these changes. Dr. Jennifer Pollock, has extensive experience with all of the biomarker assays including ET-1. Dr. Pollock runs bio-analytical core labs for two PO1s and has published extensively on these and similar methods in human and animal samples.

Additional rationale for this project is based on recent 24-hour urine results for creatinine clearance and total protein excretion from 97 patients with sickle cell anemia (Hb SS) and sickle beta zero thalassemia (SB0-thalassemia) followed in the Augusta Sickle Cell Clinic. These patients ranged in age from 19-63 years (52 females, 45 males). Of these, 17 (18%) had microalbuminuria as defined by a 24-hour albumin excretion of 150-300 mg, 34 (36%) had macroalbuminuria (>300 mg albumin excretion/24-hours), thus 54% of the patients had microalbuminuria or macroalbuminuria and only 46% were normo albuminuric. 58 patients (58%) were on chronic hydroxyurea therapy. 9 patients were on angiotensin converting enzyme inhibitors (ACEi) and 20 were on angiotensin receptor blockers (ARBs) (total 30%). 55 patients (57%) had glomerular hyperfiltration (creatinine clearance of >120 ml/min). There was an age related decline in the glomerular filtration rate (GFR) observed. The number of patients with normo albuminuria shows a sharp decline by age indicative of the progression of sickle nephropathy. Recent studies of pain in SCD have led to a change in perception. Approximately 50% of the patients reported experiencing daily, chronic pain. In addition, issues related to centralization and neuropathic pain in this patient population has begun to gain increasing attention. A large body of evidence suggests that endothelin-1 plays an important role in enhancing pain stimuli and nociception in various conditions. This is mediated by ETA receptor. Berkeley SCD transgenic mice do have hyperalgesia as shown in the rationale preliminary data section of Aim 2 and ETA receptor blockade reverses this hyperalgesia towards normal. As part of an ongoing National Institute on Minority Health and Health Disparities (NIMHD) funded study of pain and its genetic correlates (study reference: 1 P20 MD003383-01), the investigators have found that SCD patients display significant hyperalgesia as measured by pressure pain algometer testing. The testing was done at three different anatomic sites in patients (n=38) and controls (n=20) and showed that SCD patients perceived pain at significantly lower pressures compared to controls (masseter: 157.7 kilopascal (kPa) for patients, 214.4 kPa for controls, p=0.017; ulna: 299.1 kPa for patients, 477.5 kPa for controls, p=0.0018; and trapezius: 290.1 kPa for patients, 462.8 kPa for controls, p=0.02). These data suggest that hyperalgesia is present in the vast majority of SCD patients and will constitute an objective parameter to monitor during the study.

Protocol-required assessments performed at every study visit include: physical exam, vital signs, con medication review, study drug accountability, adverse events review, pain diary completion, and pregnancy testing if applicable.

Protocol-required assessments performed at specified study visits include: collection of blood and urine for safety and efficacy testing; electrocardiogram (ECG); echocardiogram (echo); Quantitative Sensory Testing (pressure pain threshold via algometer, cutaneous mechanical pain via monofilament, and thermal testing via Q-Sense Small Fiber Test); transcranial Doppler (TCD); forearm blood flow measurement; skin blood flow measurement; and completion of quality of life questionnaires.

Description of Procedures:

Sensory Testing: Patients will also undergo sensory testing at baseline and at the end of the study period. Sensory testing will include: 1) Pressure pain threshold will be measured by a hand-held, digital algometer as described by Fillingim et al at three different anatomical sites: center of right upper trapezius, right masseter, and the right ulna; 2) Cutaneous mechanical pain testing- Assessment of temporal summation of mechanical pain will be done using nylon monofilaments tested on the dorsum of the hand.; and 3) Thermal sensory testing will be performed using Q-Sense Small Fiber Test, which offers a scientifically validated measure of warm, cool and heat-pain thermal sensory thresholds.

Pain Diaries/Questionnaires: Patients will be asked to complete a daily pain diary as described in the PISCES study. The evaluation of pain diaries will be performed by Dr. Robert Gibson and the research staff. In addition, investigators will also incorporate two pre/post measures that will examine the effects of pain on functional performance and quality of life. The Assessment of Motor and Process Skills (AMPS) is a well-established functional assessment. This assessment has demonstrated the ability to discriminate between healthy controls and those with wide spread chronic pain. It also demonstrates the ability to measure change following intervention. The investigators will also measure patient's quality of life with the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me). This quality of life assessment has been specifically developed for sickle cell populations. Dr. Robert Gibson has training and experience with the ASCQ-Me and is certified to administer the AMPS.

Echocardiogram for tricuspid regurgitation jet (TRJ) Velocity Measurement: A transthoracic echocardiogram for the measurement of TRJ velocity and pulmonary artery systolic pressure will be performed at baseline (unless obtained clinically within 6 months of Day 1) and at the end of the study.

Electrocardiogram: An electrocardiogram (ECG) is a test that measures the electrical activity of the heart. An ECG will be done as a safety measure at baseline, Day 8 visit, and end of study, although ambrisentan is not known to prolong corrected QT interval (QTc).

Forearm Blood Flow Measurement: Brachial artery flow-mediated dilation (FMD) will be performed in accordance to the recent tutorial for ultrasound assessment of FMD. Patients will be tested under fasting conditions in a controlled environment at baseline and at the end of the study period.

Skin Blood Flow Measurement: Skin blood flow will be measured non-invasively using a low frequency laser imaging camera and/or a small skin probe. Ring-shaped probes that are about 1.5 inches wide will be placed on the forearm with sticky tape. One ring will be filled with approximately 2 ml (about 1/2 teaspoon) of water for local heat and the others will be used for iontophoresis. For local heat, investigators will heat the water in the ring to between 42°C (107°F) and 44°C (111°F) and wait approximately 30 minutes for the increase in skin blood flow to become stable. Iontophoresis is a technique that delivers a vasoactive drug about 1 mm deep into the skin using a low level electrical current. The advantage of this technique is that it is non-invasive and the drug does not go into the body, it just remains at the surface of the skin. We will use a 1-2% solution of either acetylcholine, sodium nitroprusside, or N-nitro-L-arginine methyl ester (L-NAME) (vasoactive substances) to increase or decrease skin blood flow. Multiple short currents (10-180 seconds) will be performed approximately 1 minute apart. Investigators will monitor skin blood flow through the ring during the forearm arterial blood flow test described above as well as during local heat and iontophoresis.

Blood and Urine Measurement: Lab tests to be performed for safety/ efficacy assessments at specified study visits include complete blood count (CBC), complete metabolic panel (CMP), spot urine for albumin-creatinine ratio, 24-hour urine, pregnancy testing, biomarkers, and inflammatory markers.

Transcranial Doppler (TCD): Pre- and post-treatment TCD will be performed to assess velocity of cerebral blood flow. This non-invasive test is performed while the subject is lying down and involves use of sound waves to assess macro-circulation in the head. A transducer is used to hear and record the results.

ELIGIBILITY:
Inclusion Criteria:

1. SS or Sβo-thalassemia
2. Age 18-65 years
3. Microalbuminuria (24-hour albumin 150-300 mg) or macroalbuminuria (24-hour albumin >300 mq) OR random urine albumin-creatinine ratio (MA Random) ≥ 30 µg/ mg creatinine
4. Subjects can have Stage 1, II, or III chronic kidney disease (CKD)
5. Subjects can be on hydroxyurea, ACE inhibitors (ACEi), or angiotensin receptor blockers (ARBs) for a period of 3 months or greater
6. Females of child bearing potential must agree to use two forms of birth control with one being a barrier method; abstinence is an acceptable form of birth control

Exclusion Criteria:

1. Other genotypes of SCD
2. History of renal transplant
3. Chronic kidney disease (Stage IV and V including patients on hemo dialysis or peritoneal dialysis)
4. Patients on chronic transfusion therapy
5. Uncontrolled/poorly controlled hypertension or history of hypertension pre-dating proteinuria or
6. Known history of HIV, Hepatitis C, and/or diabetes
7. Peripheral edema
8. History of congestive heart failure or pulmonary edema
9. Recent history of coronary artery disease
10. Pregnant or breast feeding
11. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) >3-fold upper limit of normal
12. Albumin <2.5 gm/dl
13. Hemoglobin < 6 gm/dL
14. History of non-compliance with medications and clinic visits; or Inability to give informed consent; or Patient deemed ineligible or unsuitable in the judgment of investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of ambrisentan in patients with sickle cell disease measured by physical exam, vital signs, blood and urine testing, ECG (specified visits), concomitant medication review, adverse events review | Day 1 (Baseline) through Day 113

SECONDARY OUTCOMES:
Efficacy of ambrisentan in improving kidney function in patients with sickle cell disease measured by blood | Day 1 (Baseline), Day 15, Day 29, Day 57, Day 85, and Day 113
  measured by blood
Efficacy of ambrisentan in decreasing TRJ velocity | Day 1 (Baseline) and at the end of the 12 week treatment period
  measured by echocardiogram
Efficacy of ambrisentan in decreasing inflammation | Day 1 (Baseline) through Day 113
  measurement of inflammatory markers in blood
Efficacy of ambrisentan in improving micro-circulation | Day 1 (Baseline) and at the end of the 12 week treatment period
  measured by forearm and skin blood flow measurements
Efficacy of ambrisentan in improving macro-circulation | Day 1 (Baseline), and at the end of the 12 week treatment period
  measured by Transcranial Doppler (TCD)
Efficacy of ambrisentan in improving nociception/pain | Day 1 (Baseline), and at the end of the 12 week treatment period
  performance of quantitative sensory testing
Efficacy of ambrisentan in improving kidney function in patients with sickle cell disease measured by urine testing for microalbuminuria/proteinuria | Day 1 (Baseline), Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, and Day 113
  measured by urine testing for microalbuminuria/proteinuria
Efficacy of ambrisentan in improving nociception/pain | Day 1 (Baseline) through the 12 week treatment period
  assessment of pain diaries/questionnaires
Efficacy of ambrisentan in improving nociception/pain | Day 1 (Baseline) through the 12 week treatment period
  assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Kutlar, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256